CLINICAL TRIAL: NCT02499367
Title: Adaptive Phase II Randomized Non-comparative Trial of Nivolumab After Induction Treatment in Triple-negative Breast Cancer (TNBC) Patients: TONIC-trial
Brief Title: Nivolumab After Induction Treatment in Triple-negative Breast Cancer (TNBC) Patients
Acronym: TONIC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N15TON
Record Dates: First submitted 2015-07-06; First posted 2015-07-16 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
Keywords: triple negative; metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Nivolumab; Radiotherapy; Doxorubicin; Cyclophosphamide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Radiation therapy (Active Comparator): Radiotherapy on metastatic lesion
  Interventions: Drug: Nivolumab; Radiation: Radiation therapy
- Low dose doxorubicin (Active Comparator): 15mg flat dose, once weekly for 2 weeks
  Interventions: Drug: Nivolumab; Drug: Low dose doxorubicin
- Cyclophosphamide (Active Comparator): metronomic schedule, 50mg daily orally for 2 weeks
  Interventions: Drug: Nivolumab; Drug: Cyclophosphamide
- Cisplatin (Active Comparator): 40mg/m2, weekly for 2 weeks
  Interventions: Drug: Nivolumab; Drug: Cisplatin
- No induction treatment (Active Comparator)
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — nivolumab 3 mg/kg, every 2 weeks after induction treatment
Radiation: Radiation therapy — 20 Gy to metastatic lesion
  Arms: Radiation therapy
Drug: Low dose doxorubicin — 15 mg flat dose, once weekly for 2 weeks
  Arms: Low dose doxorubicin
Drug: Cyclophosphamide — metronomic schedule, 50 mg daily orally for 2 weeks
  Arms: Cyclophosphamide
Drug: Cisplatin — 40 mg/m2, weekly for 2 weeks
  Arms: Cisplatin

SUMMARY:
This is a single center non-blinded randomized non-comparative phase II trial. The first stage of the trial consists of five arms ( with induction treatment followed by nivolumab, 1 with no induction treatment before nivolumab).

For the second stage, the number of arms will be reduced based on the results obtained in the first stage.

DETAILED DESCRIPTION:
Triple negative breast cancer (TNBC) patients have a relatively high relapse rate and upon relapse the median overall survival is less than a year. No targeted therapies are currently available for this subgroup. Compared to other breast cancer subtypes, the percentage of tumor-infiltrating lymphocytes (TILs) is significantly higher in TNBC. Given the durable responses induced by the immune checkpoint inhibitor nivolumab in other advanced solid cancers, immunotherapeutic approaches, such as blockade of PD-1 by nivolumab may be the key to treat TNBC. Moreover, since classical anticancer agents can stimulate immune effector cells, the investigators hypothesize that short-term induction treatment with radiation, doxorubicin, cyclophosphamide or cisplatin induces an anticancer immune response resulting in synergistic activity with nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic triple negative breast cancer with confirmation of Estrogen Receptor (ER) and HER2 negativity on a histological biopsy of a metastatic lesion
* 18 years or older
* Metastatic lesion accessible for histological biopsy (Mandatory biopsies: pre-induction treatment, post-induction treatment, 6-weeks. Optional biopsies: 12-weeks, at progression, of irradiated site). The pre-induction treatment biopsy has to contain sufficient tumor content (≥100 tumor cells); subjects with samples that have insufficient tumor content will require re-biopsy prior to induction treatment. Interval between last treatment and pre-induction biopsy has to be at least 14 days
* One, two or three line(s) of chemotherapy for metastatic disease and with progression of disease on last treatment regimen
* Evaluable disease according to RECIST 1.1
* Metastatic lesion accessible for radiation with 1x20 Gray or 3x8 Gray
* Subjects with brain metastases are eligible if these are not symptomatic. Subjects who received prior treatment for brain metastases should be free of progression on magnetic resonance imaging (MRI) for at least 4 weeks after treatment is completed and prior to first dose of study drug administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
* WHO performance status of 0 or 1
* Adequate bone marrow function
* Adequate hepatic function
* Adequate renal function
* Signed written informed consent

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris.
* known history of leptomeningeal disease localization
* history of having received other anticancer therapies within 2 weeks of start of the study drug
* history of immunodeficiency, autoimmune disease, conditions requiring immunosuppression (>10 mgl daily prednisone equivalents) or chronic infections.
* prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody
* live vaccine within 30 days of planned start of study therapy.
* active other cancer
* positive test for hepatitis B surface virus surface antigen (HBsAg) or hepatitis
* history of uncontrolled serious medical or psychiatric illness
* any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* current pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2015-08; Primary Completion 2023-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | assessed monthly until progression; median 12 months
  Time from randomization todate of first tumor progression

SECONDARY OUTCOMES:
Overall response rate | At 12 weeks and 6 months
  complete response or partial response at 12 weeks and 6 months
Clinical benefit rate | At 6 months
  Beneficial response (complete response, partial response or stable disease) at 6 months
Toxicity of all study regimens | assessed until 100 days after of treatment end
  adverse events will be graded according to NCI Common Toxicity Criteria v 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Marleen Kok, MD, Principal Investigator — Antoni van Leeuwenhoek
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, Netherlands

REFERENCES:
- [Derived] Lin AY, Isaeva OI, Deger T, Geurts VCM, Vessies DCL, Voorwerk L, Slagter M, Moore KS, van der Leest P, Martens JWM, van den Broek D, Wessels LFA, Kok M. CfDNA-based copy-number dynamics during anti-PD1 treatment in metastatic triple negative breast cancer. Cell Rep Med. 2025 Dec 16;6(12):102512. doi: 10.1016/j.xcrm.2025.102512. PMID 41406937